CLINICAL TRIAL: NCT07030062
Title: Transcatheter Aortic Valve Replacement With Echocardiography Guidance
Brief Title: Echocardiography Guided TAVR (Echo TAVR)
Status: Recruiting | Type: Observational
Sponsor: Pan Xiangbin (Other)
Responsible Party: Sponsor-Investigator, Pan Xiangbin, Principle Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Other Study IDs: 2025-2621
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Transcatheter Aortic Valve Replacemen; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Conventional transcatheter aortic valve replacement (TAVR) relies on fluoroscopic and contrast agents. However, in high-risk patients, exposure to ionizing radiation and contrast agents is contraindicated and undesirable. Echocardiography guidance TAVR can offer a feasible and safer strategy for TAVR.

ELIGIBILITY:
Inclusion Criteria:

1. symptomatic severe AS determined by echocardiography and Doppler that requiring aortic valve replacement, which is defined as: mean gradient ≥40 mmHg, peak aortic velocity ≥4 m/s, and aortic valve area (AVA) ≤1 cm2 (or an indexed AVA ≤0.6 cm2/m2);
2. a history of malignancy or a high familial risk of cancer, with refusal to undergo contrast- or radiation-guided procedures;
3. chronic kidney disease and refuse to receive contrast agents or radiation exposure.

Exclusion Criteria:

Required hybrid procedures or concomitant interventions on other cardiac malformations; Deemed inoperable due to extremely high surgical risk or severe comorbidities; Had untreated clinically significant coronary vascular disease amenable to revascularization; Previously undergone aortic valve replacement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients included those with symptomatic severe aortic stenosis confirmed by echocardiography (mean gradient ≥40 mmHg, peak velocity ≥4 m/s, and AVA ≤1 cm² or indexed AVA ≤0.6 cm²/m²), individuals with a history or strong family history of cancer who refused contrast- or radiation-guided procedures, and patients with chronic kidney disease unwilling to receive contrast agents or radiation exposure. Patients were excluded if they required hybrid procedures or other cardiac interventions, were deemed inoperable due to extremely high surgical risk or severe comorbidities, had untreated significant coronary artery disease suitable for revascularization, or had previously undergone aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Valve Academic Research Consortium-3 (VARC-3) | 30-day after surgery
  VARC3 include but not limited to Mortality (all-cause and cardiovascular) Stroke and transient ischemic attack (TIA) Acute kidney injury Conduction disturbances and permanent pacemaker implantation Bleeding (updated using BARC criteria) Myocardial infarction Vascular access complications Endocarditis

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided